CLINICAL TRIAL: NCT06232226
Title: Addictions and Attention Deficit Disorder With or Without Hyperactivity
Brief Title: Attention Deficit Hyperactivity Disorder
Acronym: ADA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC23_0074
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-04

CONDITIONS: Attention Deficit Hyperactivity Disorder; Behavior Hyperactive; Behavior Disorders
Keywords: Attention Deficit Disorder with Hyperactivity; Addictive disorders; Neuropsychology; Methylphenidate; Atomoxetine; Functional impairment; Symptoms
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuropsychological assessment (Other): Determination of the neuropsychological profile
  Interventions: Other: Patients suffering from the co-occurrence of ADHD and addiction(s)

INTERVENTIONS:
Other: Patients suffering from the co-occurrence of ADHD and addiction(s) — All eligible patients over 15 years and 3 months (age limit between child psychiatry and adult psychiatry), presenting both a diagnosis of ADHD and a diagnosis of at least one addictive disorder (SUD, AUD (Alcohol Use Disorder) and/ or behavioral addiction), starting care in one of the three participating centers, and meeting the indication for treatment with MPH according to European recommendations (J. J. S. Kooij et al., 2019)

SUMMARY:
The ADA cohort aims for the systematic and standardized collection of sociodemographic, clinical and neuropsychological data, during 2 visits (inclusion and 12 months), from patients suffering from the co-occurrence of ADHD (Attention Deficit Hyperactivity Disorder) and addiction(s), in addition to the treatment as usual adapted to each situation.

DETAILED DESCRIPTION:
Information on the study and diagnosis of ADHD will be carried out during a medical evaluation consultation, as part of routine care.

The two research visits (inclusion and at 12 months) will be added by the research and will each include:

* A structured clinical interview with a research professional (traceability of oral consent, administration of structured interviews, collection of self-questionnaires, collection of care from the medical record)
* A neuropsychological assessment with a neuropsychologist

ELIGIBILITY:
Inclusion Criteria :

* Patients aged over 15 years and 3 months
* For whom a diagnosis of ADHD has been confirmed less than 6 weeks ago
* For whom the diagnosis of one or more addictive disorder(s) (substance use disorder or behavioral addiction) has been confirmed
* Meeting the indication for treatment with MPH according to European recommendations (Kooij et al., 2019)
* For patients who can actually benefit from MPH: who have not yet started taking MPH
* Social security affiliates

Exclusion Criteria :

* Presenting disorders of higher cognitive functions (at the discretion of the referring clinician or the investigator making the inclusion), making data collection impossible
* Presenting difficulties in reading or writing the French language making data collection impossible
* Unable to commit to being available for the 2 visits planned as part of the cohort
* Under guardianship or legal protection

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Functional impairment | Inclusion and 12-month follow-up
  Weiss Functional Impairment Rating Scale (WFIRS-S) (scores of the 7 domains and total score)

SECONDARY OUTCOMES:
Type and severity of ADHD | Inclusion
  Diagnostiscal Interview Voor Attention deficit hyperactivity disorder (DIVA-5)
Symptoms of ADHD | Inclusion and 12-month follow-up
  Adult ADHD Self-Report Scale Symptom Checklist (ASRS-1.1) (inattention and hyperactivity/impulsivity scores)
Addictive disorders - substance use disorders (including tobacco, alcohol and other substances) | Inclusion and 12-month follow-up
  Mini International Neuropsychiatric Interview- Simplified for Diagnostic and Statistical Manual (DSM)-5 (MINI-S)
Addictive disorders - gambling disorder | Inclusion and 12-month follow-up
  National Opinion research center DSM Screen for gambling problems (NODS)
Addictive disorders - sex addiction | Inclusion and 12-month follow-up
  Structured interview adapted from the NODS to explore the diagnostic criteria proposed by Carnes et al in 2012
Addictive disorders - gambling disorder | Inclusion and 12-month follow-up
  Structured interview adapted from the NODS to explore the diagnostic criteria proposed in the third section of the DSM-5 for the Internet gaming disorder
Addictive disorders - eating addiction | Inclusion and 12-month follow-up
  Yale Food Addiction Scale (YFAS 2.0)
Psychiatric disorders | Inclusion and 12-month follow-up
  MINI-S
Neuropsychological profile - selective attention | Inclusion and 12-month follow-up
  D2-R test (CCT standard score, E% standard score and CC standard score)
Neuropsychological profile - short-term and working memory | Inclusion and 12-month follow-up
  Digit memory test (standardized scores of numbers of items correctly recalled (direct order, indirect order, ascending order, total), span sizes (direct order, indirect order, ascending order))
Neuropsychological profile - inhibition | Inclusion and 12-month follow-up
  Stroop test (standardized execution times (naming condition, interference condition), standardized numbers of uncorrected errors (naming condition, interference condition), and standardized interference score)
Neuropsychological profile - spontaneous flexibility | Inclusion and 12-month follow-up
  Verbal fluency test (standardized scores for the number of words cited and the number of errors, in both conditions (literal and categorical))
Neuropsychological profile - planning | Inclusion and 12-month follow-up
  Zoo test (total profile score)
Psychopathological profile - impulsivity | Inclusion and 12-month follow-up
  Urgency, Premeditation (lack of), Perseverance (lack of), Sensation seeking impulsivity behavior scale (UPPS-P) (5 scores)
Psychopathological profile - emotional dysregulation | Inclusion and 12-month follow-up
  Difficulties in Emotion Regulation Scale (DERS-16) (5 scores and total score)
Psychopathological profile - sensorial profile | Inclusion and 12-month follow-up
  Sensory profile of Winnie Dunn - adult version (category and raw scores in the 4 quadrants)
Psychopathological profile - self-esteem | Inclusion and 12-month follow-up
  Rosenberg Self-Esteem Scale (RSES) (total score)
Quality of life survey | Inclusion and 12-month follow-up
  World Health Organization Quality Of Life (WHOQoL-26) (4 scores)
Care received | 12-month follow-up
  Effective implementation of treatment with MPH (yes/no) or atomoxetine (yes/no), If no, reasons for not implementing it (for MPH), Care provided (Cognitive remediation / behavioral and cognitive therapy / psychoeducation / other psychosocial intervention (details) / other drug treatment), Reported compliance and misuse for MPH and atomoxetine, Reported compliance for non-drug care, Tolerance: numerical scale from 0 to 10 for the evaluation of the main adverse effects (for MPH and for atomoxetine).
Personal and family medical history | Inclusion
  List of somatic, psychiatric and addictive disorders for personal history, list of psychiatric and addictive disorders for family history
Sociodemographics | Inclusion
  Age, gender, level of education, professional status, number of children

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Nantes University Hospital, Nantes, Loire-Atlantique
  - CHRU de Brest, Brest
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No